CLINICAL TRIAL: NCT04969055
Title: Prevalence, Clinical Features and Risk Factors of Cirrhotic Cardiomyopathy Assessed by Two-dimensional Speckle Tracking Imaging
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-qilu
Record Dates: First submitted 2021-07-11; First posted 2021-07-20 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2021-07

CONDITIONS: Liver Cirrhosis; Cirrhotic Cardiomyopathy
Keywords: Cirrhosis; cardiac dysfunction;Cardiac Imaging
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with liver cirrhosis: cirrhosis based on either clinical/radiological parameters or liver histology
  Interventions: Other: Not
- control group: Healthy ubjects without known heart disease

INTERVENTIONS:
Other: Not — Not
  Groups: patients with liver cirrhosis

SUMMARY:
The purpose of this study is to assess the prevalence of cirrhotic cardiomyopathy in patients with cirrhosis, and to analyze the correlation between the severity of cirrhosis and cardiac dysfunction. To investigate the risk factors for cirrhotic cardiomyopathy, and raise clinicians' awareness of cirrhotic cardiomyopathy, early assessment and intervention to improve long-term outcomes in patients with cirrhosis.

DETAILED DESCRIPTION:
Liver cirrhosis is the terminal stage of the development of chronic liver disease caused by various reasons, and it is often accompanied by multiple complications. Late cirrhosis is often accompanied by obvious changes in liver and systemic hemodynamics. Patients with liver cirrhosis are in a highly dynamic cycle Status: lower arterial blood pressure, increased heart rate, increased cardiac output, peripheral vascular resistance, which often lead to changes in myocardial structure and function, called cirrhotic cardiomyopathy. Cirrhotic cardiomyopathy (CCM) is defined as cardiac dysfunction in patients with end-stage liver disease in the absence of prior heart disease. The true burden of CCM among patients with ESLD is currently unknown. Prior studies evaluated CCM prevalence and estimated it to be approximately 50%, however, this estimate was based on the old criteria. In 2020, the Cirrhotic Cardiomyopathy Association updated the diagnostic criteria for cirrhotic cardiomyopathy. At present, the true prevalence of cirrhotic cardiomyopathy still needs to be reassessed. In addition, studies on the risk factors for cirrhotic cardiomyopathy are rare. Based on the above research background, carry out this research.

ELIGIBILITY:
Inclusion Criteria:

* The clear diagnosis of cirrhosis in patients caused by various reasons

Exclusion Criteria:

* History of cardiovascular disease
* Diabetes
* High blood pressure
* Hepatocellular carcinoma (HCC) or other malignant tumors
* Patients with the chronic obstructive pulmonary disease
* Thyroid diseases
* Severe infection in the last 2 weeks
* History of liver transplantation and/or TIPS surgery
* Presence of stage 3 or above chronic kidney disease or acute chronic kidney disease
* Pregnant women
* Did not sign the informed consent form and refused to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From December 1, 2020 to December 31, 2021, The clear diagnosis of cirrhosis in patients caused by various reasons who have come to our hospital for digestive medicine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
cirrhotic cardiomyopathy | Within 48 hours after hospitalization
  Different levels of left ventricular diastolic dysfunction in patients with liver cirrhosis

OTHER OUTCOMES:
N-terminal Pro-brain Natriuretic Peptide serum level | Within 48 hours after hospitalization
  Venous blood sampling was performed in the morning, after a 12-h fast. serum levels of NT-proBNP were measured by an electrochemiluminescence immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: YanJing Gao, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital , Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Xu H, Zhang Y, Gao Y. Prevalence and risk factors for cirrhotic cardiomyopathy: a prospective cross-sectional study. Eur J Gastroenterol Hepatol. 2024 Apr 1;36(4):469-475. doi: 10.1097/MEG.0000000000002716. Epub 2024 Feb 16. PMID 38407871